CLINICAL TRIAL: NCT04586790
Title: The Effect of Oral Midodrine Versus Oral Desmopressin Acetate Use for Liberation From IV Noradrenaline in Intensive Care Unit Patients Recovering From Spinal Shock .
Brief Title: the Effect of Oral Vasopressors for Liberation From IV Vasopressors in Spinal Shock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed talaat ahmed aly (Other)
Responsible Party: Sponsor-Investigator, Ahmed talaat ahmed aly, clinical professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oral vasopressors
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Spinal Shock
MeSH Terms: interventions — Midodrine; Deamino Arginine Vasopressin; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- midodrine group (Experimental): midodrine group will receive midodrine 10 mg PO q8hr with gradual weaning of IV noradrenaline after receiving 4 doses of oral midodrine
  Interventions: Drug: Midodrine Oral Tablet
- minirin group (Experimental): the patients will receive minirin 60 µg PO q8hr with gradual weaning of IV noradrenaline after receiving 4 doses of oral minirin
  Interventions: Drug: Minirin oral tablet
- control group (Experimental): the patients will receive IV nor-adrenaline and are gradually weaning from it according to routine hospital care without adding oral midodrine or oral minirin .
  Interventions: Drug: Nor-Adrenaline

INTERVENTIONS:
Drug: Midodrine Oral Tablet — midodrine group will receive midodrine 10 mg PO q 8 hr with gradual weaning of IV nor-adrenaline after receiving 4 doses of oral midodrine .
  Arms: midodrine group
Drug: Minirin oral tablet — Minirin group will receive minirin 60 µg PO q 8 hr with gradual weaning of IV nor-adrenaline after receiving 4 doses of oral minirin .
  Arms: minirin group
Drug: Nor-Adrenaline — control group will receive IV nor-adrenaline and is gradually weaning from it according to routine hospital care without adding oral midodrine or oral minirin .
  Arms: control group

SUMMARY:
the study is developed to evaluate the effect of use of oral vasopressors (midodrine versus minirin) on weaning ICU patients from IV vasopressors (noradrenaline) and compare between them for efficacy in shortage the duration of IV vasopressor and has low complications and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* Patients of both genders.
* Patients diagnosed by spinal shock and they are in the recovery stage .

Exclusion Criteria:

* Patient refusal.
* Anuric or oliguric patients or patients with chronic kidney disease.
* Patients with allergy to medication included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-28 (Estimated)

PRIMARY OUTCOMES:
liberation the patient from IV vasopressors with maintaining hemodynamics. | 48 hrs
  Blood pressure will be assessed regularly every 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Ahmed, lecture, Principal Investigator — Assiut University
Locations (1):
- Ahmed Talaat Ahmed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No